CLINICAL TRIAL: NCT03918187
Title: Nalbuphine Versus Midazolam as an Adjuvant to Intrathecal Bupivacaine for Postoperative Analgesia in Patients Undergoing Cesarean Section
Brief Title: Intrathecal Nalbuphine Versus Midazolam in Cesarean Section
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, olfat abd elmoniem ibrahem, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5305
Record Dates: First submitted 2019-04-07; First posted 2019-04-17 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Cesarean Section Pain
Keywords: nalbuphine; midazolam
MeSH Terms: interventions — Bupivacaine; Nalbuphine; Midazolam

STUDY DESIGN:
Intervention Model Description: Controlled comparative Double blind randomized study
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bupivacaine (Experimental): 12.5 mg hyperbaric bupivacaine + 0.5 ml 0.9% normal saline .
  Interventions: Drug: Bupivacaine
- nalbuphine (Active Comparator): 12.5 mg hyperbaric bupivacaine + 1 mg nalbuphine add in 0.5 ml 0.9% normal saline.
  Interventions: Drug: Nalbuphine
- midazolam (Active Comparator): 12.5 mg hyperbaric bupivacaine + 2.5 mg midazolam .
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Bupivacaine — compare between nalbuphine versus midazolam as an adjuvant to intrathecal bupivacain to evaluate postoperative analgesia .
  Arms: bupivacaine
Drug: Nalbuphine — compare between nalbuphine versus midazolam as an adjuvant to intrathecal bupivacain to evaluate postoperative analgesia .
  Arms: nalbuphine
Drug: Midazolam — compare between nalbuphine versus midazolam as an adjuvant to intrathecal bupivacain to evaluate postoperative analgesia .
  Arms: midazolam

SUMMARY:
Adequate pain management is important to facilitate the functional recovery and enable the patients for rapid rehabilitation of normal activity .

Various adjuvants were being used with intrathecal bupivacain to prolong & improve postoperative pain relief in patients undergoing cesarean section .

The aim of this study was to compare intrathecal nalbuphine versus intrathecal midazolam in patient undergoing cesarean section. The investigators primary aims were to compare the characteristics of sensory and motor block, the effective analgesic time, and analgesic requirement. Secondary aims were to compare the side effects, sedation score and apgare score.

DETAILED DESCRIPTION:
Analgesia is the main point for each patient postoperatively. It is important to provide good analgesia with less hazardous (1). Cesarean section is a painful operation in need for adequate postoperative analgesia (1). Adequate pain management is important to facilitate the functional recovery and enable the patients for rapid rehabilitation of their normal activity (2).

Cesarean section was done under general anesthesia (GA) or regional anesthesia. The subarachnoid blockade is the preferred procedure (3). It avoids the depressant effect of GA on neonate and also the risk of aspiration, with better postoperative pain relief. However the most commonly local anesthetic used, hyperbaric bupivacaine has limited effect lasts for 1.5 - 2 hours (4). Its onset was slow with short duration of postoperative analgesia (3).

Adjuvant drugs added to bupivacaine intrathecally improve the duration and quality of the blockade and prolong the postoperative analgesia (5). Various adjuvants were being used such as alpha2 agonists, neostigmine, opiates, and ketamine etc, yet no drug was identified to specifically inhibit nociception without side effects (6).

Nalbuphine is a synthetic opioid with mixed agonist antagonist effect. It provides a significantly rapid onset of pain relief probably because of its lipophilic properties. It binds to both mu-and kappa receptors, binding of nalbuphine to mu receptors competitively displace other mu-agonists from these receptors without any agonist activity. Therefore decrease the side effects of mu agonist (nausea, vomiting, respiratory depression , urinary retention, pruritis and prolonged sedation) (7). While when binds to kappa receptors nalbuphine has agonist effect (analgesic effect) through the kappa receptors distributed in the brain and spinal cord(1). There were no documented studies of nalbuphine neurotoxicity (5, 8).

Benzodiazepines are used mainly for sedation, anoxiolysis and amnesia. Discovery of their receptors in spinal cord allow the use of midazolam intrathecally for analgesia. Several studies show that the addition of intrathecal midazolam potentiates the analgesic effect of intrathecal bupivacain without significant side effects, or neurotoxicity (9, 10).

There are several studies studied the effect of intrathecal nalbuphine and intrathecal midazolam but to The investigators knowledge no study compares between them.

The aim of this study was to compare intrathecal nalbuphine versus intrathecal midazolam in patient undergoing cesarean section. The investigators primary aims were to compare the characteristics of sensory and motor block, the effective analgesic time, and analgesic requirement. Secondary aims were to compare the side effects, sedation score and apgare score.

ELIGIBILITY:
Inclusion Criteria: -

* Female gender .
* Age : 18 - 40 years old .
* Physical status : ASA II .
* Elective cesarean section

Exclusion Criteria:

* - Patient refusal .
* History of hypertension or cardiac diseases .
* Psychiatric disorders .
* Coagulopathy .
* Allergy to study drugs .
* Contraindication to spinal anesthesia .
* Failure of spinal anesthesia .

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Effective analgesic time | up to six hours postoperative
  the time start from intrathecal injection to the first analgesic dose.
Total postoperative analgesic dose . | 24 hours
  the analgesic dose consumed
Onset of sensory and motor block | up tp five minutes after intrathecal injection
  the time of onset of sensory and motor block
duration of sensory and motor block | up to five hours postoperative
  the time of duration of sensory and motor block

SECONDARY OUTCOMES:
Sedation score | one hour during surgery
  score of sedation:
  1= awake and alert 2 = sedated ,respond to verbal stimules 3= sedated respond to a mild physical status 4=sedated respond to a moderate or strong physical stimuls 5= not arousable 5 is the higher value
Apgar score | 1-5 minutes after delivery
  score for baby
number of participants with hypotension , bradycardia ,vomiting , nausea , shivering number of participants with hypotension , bradycardia ,vomiting , nausea , shivering | up to 24 hours postoperative
  incidence of hypotension , bradycardia ,vomiting , nausea , shivering

CONTACTS AND LOCATIONS:
Overall Officials: Olfat A I Amin, MD, Principal Investigator — Zagazig University
Locations (1):
- Olfat Abd Elmoniem Ibrahem Amin, Zagazig, Eygpt/zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amin OAI, Ibrahem MA, Salem DAE. Nalbuphine versus Midazolam as an Adjuvant to Intrathecal Bupivacaine for Postoperative Analgesia in Patients Undergoing Cesarean Section. J Pain Res. 2020 Jun 11;13:1369-1376. doi: 10.2147/JPR.S242545. eCollection 2020. PMID 32606903